CLINICAL TRIAL: NCT02253654
Title: A Randomized, Multicenter, Double-blind Study Evaluating Two Epoetin Alfa Dosing Strategies in Subjects With Chronic Kidney Disease Receiving Hemodialysis
Brief Title: Evaluation of Two Epoetin Alfa Dosing Strategies in Subjects With Chronic Kidney Disease Receiving Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110208
Record Dates: First submitted 2014-09-11; First posted 2014-10-01 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Renal Insufficiency, Chronic; Anemia; Renal Dialysis; Erythrocyte Transfusion
Keywords: Chronic Kidney Disease; Anemia; Hemodialysis; Red Blood Cell Transfusion
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoetin alfa Alternative Titration (Experimental): Participants received epoetin alfa administered intravenously three times a week during hemodialysis for up to 37 weeks. For the first two weeks the dose of epoetin alfa was based on the dose at the time of screening. Beginning at week 3 dose changes may have occurred every 2 weeks according to the alternative dosing algorithm, where smaller, frequent dose adjustments were permitted based on six hemoglobin categories.
  Interventions: Drug: Epoetin alfa
- Epoetin alfa USPI Titration (Active Comparator): Participants received epoetin alfa administered intravenously three times a week during hemodialysis for 37 weeks. For the first two weeks the dose of epoetin alfa was based on the dose at the time of screening. Beginning at week 3 dose decreases were permitted every 2 weeks and beginning at week 5 dose increases could only occur ≥ 4 weeks from the last dose increase, according to the United States package insert (USPI) dosing algorithm which includes four categories of hemoglobin levels.
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — Administered intravenously (IV) three times a week (TIW) by appropriately trained healthcare professionals during hemodialysis.
  Other Names: Epogen

SUMMARY:
The purpose of this study is to compare two different dosing methods of epoetin alfa and their effectiveness in maintaining hemoglobin levels between 10.0 to 11.0 g/dL in in patients with chronic kidney disease (CKD) receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained prior to initiation of any study-specific activities/procedures
* Age 18 or older
* Prescribed hemodialysis three times a week (TIW) for ≥ 12 weeks prior to randomization
* Prescribed IV administration of epoetin alfa TIW for ≥ 12 weeks prior to randomization
* Prescribed ≥ 3000 Units/week (ie, ≥ 1000 Units/administration) and < 90,000 Units/week (ie, < 30,000 Units/administration) of epoetin alfa during the 4 weeks prior to randomization
* Received ≥ 4 doses of epoetin alfa during the 2 weeks prior to randomization
* Hemoglobin concentration ≤ 11.0 g/dL, per the most recent local laboratory value obtained during the 2 weeks prior to randomization
* Hemoglobin concentration ≤ 11.0 g/dL, at the screening visit, using the hemoglobin point of care device provided by Amgen
* Iron replete, defined as a transferrin saturation (TSAT) ≥ 20% and a ferritin ≥ 100 ng/mL, per the most recent local laboratory value obtained during the 4 weeks prior to randomization

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s) prior to randomization
* Other investigational procedures while participating in this study are excluded
* Systemic hematologic disease (eg, sickle cell anemia, myelodysplastic syndrome, hematologic malignancy)
* Current or prior malignancy within 5 years of randomization, with the exception of non-melanoma skin cancers, cervical or breast ductal carcinoma in situ
* Treatment for any malignancy (eg, radiation, chemotherapy, hormone therapy or biologics) within 5 years of randomization, with the exception of locally excised non-melanoma skin cancers, cervical or breast ductal carcinoma in situ
* Subject is currently pregnant or planning to become pregnant during treatment and for 30 days after the end of treatment
* Subject is currently breast feeding or planning on breast feeding during treatment and for 30 days after the end of treatment
* Females of reproductive potential who are not willing to use an acceptable method of effective contraception during treatment and for at least 30 days after the end of treatment
* Currently receiving IV antibiotics
* Currently receiving systemic immunosuppressive therapy known to cause anemia, including treatment for active hepatitis (eg, azathioprine, mycophenolate mofetil, ≥ 10 mg prednisone [or equivalent]/day, interferon)
* Known human immunodeficiency virus (HIV) positive
* Known neutralizing anti-erythropoietic protein antibodies
* Known sensitivity to epoetin alfa
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, planned vacations where away from dialysis unit for more than 2 weeks) to the best of the subject and investigator's knowledge
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Previously entered this study
* Occurrence of any of the following within 8 weeks prior to randomization:

  * Seizure
  * Clinically relevant active bleeding (eg, gastrointestinal bleed)
  * RBC transfusion
  * Any hospitalization or observational stay > 24 hours
* Uncontrolled hypertension, per the investigator within the 4 weeks prior to randomization
* Expected or scheduled solid organ transplant(eg, kidney) within 40 weeks after randomization
* Expected or scheduled to change dialysis modality (eg, peritoneal dialysis, home hemodialysis) within 40 weeks after randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- United States (34):
  - Research Site, Cerritos, California
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Montebello, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, Simi Valley, California
  - Research Site, Vacaville, California
  - Research Site, Whittier, California
  - Research Site, Miami, Florida
  - Research Site, Miami Gardens, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Macon, Georgia
  - Research Site, Statesboro, Georgia
  - Research Site, Merrillville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Astoria, New York
  - Research Site, Brooklyn, New York
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Carrboro, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Meadville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Hampton, Virginia
  - Research Site, Norfolk, Virginia
- Research Site, Toa Baja, Puerto Rico

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 31 centers in the United States. Participants were enrolled from 01 April 2015 to 17 August 2015.
Pre-assignment Details: Eligible participants with anemia and chronic kidney disease who were receiving hemodialysis were randomized in a 1:1 ratio to 1 of 2 dosing algorithms.
Period: Overall Study
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Started | 108 | 108
Received Treatment | 104 | 107
Completed | 85 | 90
Not Completed | 23 | 18
Not completed — Withdrawal by Subject | 12 | 4
Not completed — Decision by Sponsor | 1 | 1
Not completed — Lost to Follow-up | 2 | 5
Not completed — Death | 4 | 7
Not completed — Did Not Receive Study Treatment | 4 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration | Total
Number analyzed (Participants) | 108 | 108 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.3) | 58.7 (14.2) | 59.8 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 40 | 88
  Male | 60 | 68 | 128
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 7 | 7 | 14
  Black | 53 | 50 | 103
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 40 | 40 | 80
  Other | 8 | 10 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 30 | 39 | 69
  Not Hispanic/Latino | 78 | 69 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Hemoglobin Measurements Within 10 to 11 g/dL During the Evaluation Period
Description: Hemoglobin was measured every 2 weeks during the evaluation period. The percentage of these measurements that were within the range of 10-11 g/dL was calculated for each participant.
Time Frame: The evaluation period (weeks 13-37)
Population: The Primary Analysis Set which consists of all randomized participants who had at least 6 hemoglobin measurements during the evaluation period while on study and receiving investigational product.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin measurements
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
percentage of hemoglobin measurements | 46.41 (2.39) | 46.02 (2.56)
Statistical Analysis 1: Comparison: Epoetin Alfa Alternative Titration vs Epoetin Alfa USPI Titration; The difference between treatment groups for the percent of hemoglobin measurements within 10.0 to 11.0 g/dL during the evaluation period was tested using a 1-sided t-test with a significance level of 0.025; Test type: Superiority or Other; p = 0.46, t-test, 1 sided; Treatment difference = 0.39, 97.5% CI 1-sided [lower limit -6.58], Standard Error of Mean 3.53

2. Secondary Outcome: Hemoglobin Concentration at Each Visit
Time Frame: Baseline (screening visit) and weeks 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
Population: Primary analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
g/dL
  Baseline (n = 89, 100) | 10.15 (0.66) | 10.04 (0.81)
  Week 3 (n = 89, 100) | 10.54 (0.88) | 10.34 (0.97)
  Week 5 (n = 89, 99) | 10.66 (0.93) | 10.51 (1.04)
  Week 7 (n = 88, 97) | 10.45 (1.02) | 10.28 (1.07)
  Week 9 (n = 89, 100) | 10.32 (1.16) | 9.97 (0.87)
  Week 11 (n = 88, 99) | 10.33 (1.05) | 10.15 (0.88)
  Week 13 (n = 89, 100) | 10.28 (1.04) | 9.99 (0.91)
  Week 15 (n = 89, 100) | 10.46 (1.38) | 9.98 (0.93)
  Week 17 (n = 89, 100) | 10.20 (1.05) | 10.01 (1.22)
  Week 19 (n = 89, 100) | 10.37 (1.14) | 9.94 (0.87)
  Week 21 (n = 87, 99) | 10.33 (1.01) | 9.92 (0.81)
  Week 23 (n = 88, 98) | 10.46 (1.05) | 10.03 (0.86)
  Week 25 (n = 87, 98) | 10.56 (1.00) | 9.94 (0.97)
  Week 27 (n = 88, 94) | 10.32 (1.10) | 9.97 (0.86)
  Week 29 (n =89, 92) | 10.34 (1.01) | 10.02 (1.07)
  Week 31 (n = 85, 89) | 10.34 (0.95) | 9.96 (1.07)
  Week 33 (n = 86, 90) | 10.18 (1.00) | 10.05 (0.92)
  Week 35 (n = 87, 88) | 10.12 (1.23) | 9.94 (0.90)
  Week 37 (n = 87, 93) | 10.10 (1.11) | 9.86 (0.85)

3. Secondary Outcome: Percentage of Participants With Transfusion Events Overall and During Each Study Period
Description: The percentage of participants who received red blood cell (RBC) transfusions during the study and during each study period.
Time Frame: Overall Study: Study week 1 to week 41; Titration Period: Study week 1 to week 12; Evaluation Period: Study week 13 to week 37; Safety Follow-up Period: Study week 38 to week 41
Population: Primary analysis set with available data in each study period
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
percentage of participants
  Overall (n = 89, 100) | 6.7 | 12.0
  Titration Period (n = 89, 100) | 2.2 | 1.0
  Evaluation Period (n = 89, 100) | 5.6 | 10.0
  Safety Follow-up Period (n = 83, 90) | 1.2 | 1.1

4. Secondary Outcome: Hemoglobin Rate of Change at Each Visit
Description: Hemoglobin rate of change (ROC) was calculated for each visit using the following formula: ROC = (current visit hemoglobin value - previous visit hemoglobin value) / number of days between each visit * 14. A positive value indicates a rate of rise and a negative value indicates a rate of decline.
Time Frame: Baseline (screening visit) and weeks 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
Population: Primary analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: g/dL/2 weeks
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
g/dL/2 weeks
  Week 3 (n = 89, 100) | 0.36 (0.79) | 0.27 (0.71)
  Week 5 (n = 89, 99) | 0.10 (0.81) | 0.13 (1.01)
  Week 7 (n = 88, 97) | -0.22 (0.90) | -0.19 (1.42)
  Week 9 (n = 89, 100) | -0.12 (0.93) | -0.28 (1.08)
  Week 11 (n = 88, 99) | 0.02 (1.01) | 0.19 (0.67)
  Week 13 (n = 89, 100) | -0.05 (0.93) | -0.19 (0.97)
  Week 15 (n = 89, 100) | 0.19 (1.01) | -0.01 (0.87)
  Week 17 (n = 89, 100) | -0.22 (1.08) | 0.02 (1.07)
  Week 19 (n = 89, 100) | 0.18 (0.97) | -0.06 (1.25)
  Week 21 (n = 87, 99) | -0.02 (0.74) | -0.06 (0.72)
  Week 23 (n = 88, 98) | 0.16 (0.87) | 0.09 (0.78)
  Week 25 (n = 87, 98) | 0.07 (0.78) | -0.06 (0.84)
  Week 27 (n = 88, 94) | -0.18 (0.77) | 0.01 (0.85)
  Week 29 (n =89, 92) | 0.04 (0.86) | 0.05 (0.73)
  Week 31 (n = 85, 89) | -0.02 (0.72) | -0.03 (0.74)
  Week 33 (n = 86, 90) | -0.16 (0.82) | 0.06 (0.74)
  Week 35 (n = 87, 88) | -0.05 (0.98) | -0.13 (0.72)
  Week 37 (n = 87, 93) | -0.04 (1.00) | -0.03 (0.64)

5. Secondary Outcome: Hemoglobin Intra-subject Variability
Description: Intra-subject variability was defined for each participant as the standard deviation (SD) of all of the hemoglobin concentrations during the evaluation period for the participant. The mean intra-subject SD for all participants is the sum of the intra-subject SDs divided by the total number of participants evaluated.
Time Frame: The evaluation period (weeks 13 to 37)
Population: Primary analysis set
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
g/dL | 0.74 (0.30) | 0.70 (0.32)

6. Secondary Outcome: Percentage of Participants With Hemoglobin Excursions at Each Visit
Description: An excursion is identified as an event when a hemoglobin concentration fell below or exceeded the pre-specified thresholds of: - < 9.0 g/dL, or - > 11.0 g/dL, or - > 12.0 g/dL. The percentage of participants with any excursions and excursions in each subcategory at each time point and overall during the study are reported.
Time Frame: Baseline (screening visit) and weeks 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, and 37
Population: Primary analysis set with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
percentage of participants
  Overall Excursions (n = 89, 100) | 91.0 | 93.0
  Overall Excursions < 9.0 (n = 89, 100) | 48.3 | 61.0
  Overall Excursions > 11.0 (n = 89, 100) | 80.9 | 83.0
  Overall Excursions > 12.0 (n = 89, 100) | 25.8 | 19.0
  Baseline Excursions (n = 89, 100) | 3.4 | 11.0
  Baseline Excursions < 9.0 (n = 89, 100) | 3.4 | 11.0
  Baseline Excursions > 11.0 (n = 89, 100) | 0.0 | 0.0
  Baseline Excursions > 12.0 (n = 89, 100) | 0.0 | 0.0
  Week 3 Excursions (n = 89, 100) | 29.2 | 27.0
  Week 3 Excursions < 9.0 (n = 89, 100) | 2.2 | 6.0
  Week 3 Excursions > 11.0 (n = 89, 100) | 27.0 | 21.0
  Week 3 Excursions > 12.0 (n = 89, 100) | 5.6 | 5.0
  Week 5 Excursions (n = 89, 99) | 36.0 | 29.3
  Week 5 Excursions < 9.0 (n = 89, 99) | 1.1 | 4.0
  Week 5 Excursions > 11.0 (n = 89, 99) | 34.8 | 25.3
  Week 5 Excursions > 12.0 (n = 89, 99) | 5.6 | 7.1
  Week 7 Excursions (n = 88, 97) | 27.3 | 28.9
  Week 7 Excursions < 9.0 (n = 88, 97) | 6.8 | 8.2
  Week 7 Excursions > 11.0 (n = 88, 97) | 20.5 | 20.6
  Week 7 Excursions > 12.0 (n = 88, 97) | 3.4 | 4.1
  Week 9 Excursions (n = 89, 100) | 29.2 | 17.0
  Week 9 Excursions < 9.0 (n = 89, 100) | 9.0 | 10.0
  Week 9 Excursions > 11.0 (n = 89, 100) | 20.2 | 7.0
  Week 9 Excursions > 12.0 (n = 89, 100) | 3.4 | 0.0
  Week 11 Excursions (n = 88, 99) | 22.7 | 23.2
  Week 11 Excursions < 9.0 (n = 88, 99) | 4.5 | 7.1
  Week 11 Excursions > 11.0 (n = 88, 99) | 18.2 | 16.2
  Week 11 Excursions > 12.0 (n = 88, 99) | 2.3 | 1.0
  Week 13 Excursions (n = 89, 100) | 25.8 | 21.0
  Week 13 Excursions < 9.0 (n = 89, 100) | 7.9 | 9.0
  Week 13 Excursions > 11.0 (n = 89, 100) | 18.0 | 12.0
  Week 13 Excursions > 12.0 (n = 89, 100) | 4.5 | 1.0
  Week 15 Excursions (n = 89, 100) | 27.0 | 24.0
  Week 15 Excursions < 9.0 (n = 89, 100) | 5.6 | 13.0
  Week 15 Excursions > 11.0 (n = 89, 100) | 21.3 | 11.0
  Week 15 Excursions > 12.0 (n = 89, 100) | 6.7 | 0.0
  Week 17 Excursions (n = 89, 100) | 23.6 | 21.0
  Week 17 Excursions < 9.0 (n = 89, 100) | 9.0 | 12.0
  Week 17 Excursions > 11.0 (n = 89, 100) | 14.6 | 9.0
  Week 17 Excursions > 12.0 (n = 89, 100) | 4.5 | 3.0
  Week 19 Excursions (n = 89, 100) | 28.1 | 19.0
  Week 19 Excursions < 9.0 (n = 89, 100) | 9.0 | 13.0
  Week 19 Excursions > 11.0 (n = 89, 100) | 19.1 | 6.0
  Week 19 Excursions > 12.0 (n = 89, 100) | 9.0 | 0.0
  Week 21 Excursions (n = 87, 99) | 27.6 | 17.2
  Week 21 Excursions < 9.0 (n = 87, 99) | 8.0 | 12.1
  Week 21 Excursions > 11.0 (n = 87, 99) | 19.5 | 5.1
  Week 21 Excursions > 12.0 (n = 87, 99) | 3.4 | 0.0
  Week 23 Excursions (n = 88, 98) | 29.5 | 20.4
  Week 23 Excursions < 9.0 (n = 88, 98) | 6.8 | 10.2
  Week 23 Excursions > 11.0 (n = 88, 98) | 22.7 | 10.2
  Week 23 Excursions > 12.0 (n = 88, 98) | 5.7 | 0.0
  Week 25 Excursions (n = 87, 98) | 28.7 | 20.4
  Week 25 Excursions < 9.0 (n = 87, 98) | 2.3 | 13.3
  Week 25 Excursions > 11.0 (n = 87, 98) | 26.4 | 7.1
  Week 25 Excursions > 12.0 (n = 87, 98) | 5.7 | 2.0
  Week 27 Excursions (n = 88, 94) | 29.5 | 21.3
  Week 27 Excursions < 9.0 (n = 88, 94) | 10.2 | 16.0
  Week 27 Excursions > 11.0 (n = 88, 94) | 19.3 | 5.3
  Week 27 Excursions > 12.0 (n = 88, 94) | 3.4 | 0.0
  Week 29 Excursions (n = 89, 92) | 25.8 | 29.3
  Week 29 Excursions < 9.0 (n = 89, 92) | 5.6 | 16.3
  Week 29 Excursions > 11.0 (n = 89, 92) | 20.2 | 13.0
  Week 29 Excursions > 12.0 (n = 89, 92) | 4.5 | 2.2
  Week 31 Excursions (n = 85, 89) | 20.0 | 28.1
  Week 31 Excursions < 9.0 (n = 85, 89) | 4.7 | 16.9
  Week 31 Excursions > 11.0 (n = 85, 89) | 15.3 | 11.2
  Week 31 Excursions > 12.0 (n = 85, 89) | 5.9 | 1.1
  Week 33 Excursions (n = 86, 90) | 22.1 | 22.2
  Week 33 Excursions < 9.0 (n = 86, 90) | 7.0 | 11.1
  Week 33 Excursions > 11.0 (n = 86, 90) | 15.1 | 11.1
  Week 33 Excursions > 12.0 (n = 86, 90) | 3.5 | 2.2
  Week 35 Excursions (n = 87, 88) | 26.4 | 21.6
  Week 35 Excursions < 9.0 (n = 87, 88) | 11.5 | 13.6
  Week 35 Excursions > 11.0 (n = 87, 88) | 14.9 | 8.0
  Week 35 Excursions > 12.0 (n = 87, 88) | 4.6 | 0.0
  Week 37 Excursions (n = 87, 93) | 20.7 | 17.2
  Week 37 Excursions < 9.0 (n = 87, 93) | 8.0 | 12.9
  Week 37 Excursions > 11.0 (n = 87, 93) | 12.6 | 4.3
  Week 37 Excursions > 12.0 (n = 87, 93) | 3.4 | 0.0

7. Secondary Outcome: Weekly Epoetin Alfa Dose at Each Visit
Time Frame: Weeks 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, and 35
Population: Primary analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
units
  Week 1 (n = 89, 100) | 13139.9 (9360.1) | 10400 (8439.9)
  Week 3 (n = 89, 100) | 9683.7 (9162.9) | 6912.5 (7459.4)
  Week 5 (n = 89, 100) | 8324.2 (8689.7) | 6874.0 (8204.3)
  Week 7 (n = 89, 100) | 9319.1 (7977.5) | 6411.0 (7040.6)
  Week 9 (n = 89, 100) | 9253.4 (8536.9) | 8003.0 (7292.8)
  Week 11 (n = 89, 100) | 10039.3 (9194.1) | 6483.0 (6854.9)
  Week 13 (n = 89, 100) | 10358.4 (10247.7) | 7387.5 (7271.6)
  Week 15 (n = 89, 100) | 8889.3 (8316.8) | 6874.5 (5952.9)
  Week 17 (n = 89, 100) | 10251.7 (9973.7) | 6924.5 (6211.1)
  Week 19 (n = 89, 100) | 10475.8 (10437.0) | 7112.5 (6300.4)
  Week 21 (n = 89, 99) | 9605.1 (8225.0) | 6909.6 (6102.5)
  Week 23 (n = 89, 98) | 8905.1 (7748.3) | 6830.1 (6397.0)
  Week 25 (n = 89, 98) | 7543.8 (7225.1) | 7486.7 (6676.2)
  Week 27 (n = 89, 96) | 9765.7 (12013.7) | 6662.5 (6362.8)
  Week 29 (n =89, 94) | 9088.8 (10146.9) | 6083.0 (6149.1)
  Week 31 (n = 88, 91) | 8543.2 (10821.7) | 6673.1 (6277.6)
  Week 33 (n = 87, 90) | 9019.0 (10466.9) | 6235.6 (6041.6)
  Week 35 (n = 87, 90) | 8709.2 (8631.9) | 5950.6 (5364.6)

8. Secondary Outcome: Number of RBC Units Transfused Overall and During Each Study Period
Description: The number of red blood cell (RBC) units transfused during the study and during each study period.
Time Frame: as for outcome 3
Population: Primary analysis set with available data in each study period
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Number analyzed (Participants) | 89 | 100
participants
  Overall Study: 1 RBC Unit (n = 89, 100) | 1 | 4
  Overall Study: 2 RBC Units (n = 89, 100) | 2 | 5
  Overall Study: 3 RBC Units (n = 89, 100) | 1 | 2
  Overall Study: > 3 RBC Units (n = 89, 100) | 2 | 1
  Titration Period: 1 RBC Unit (n = 89, 100) | 0 | 1
  Titration Period: 2 RBC Units (n = 89, 100) | 1 | 0
  Titration Period: 3 RBC Units (n = 89, 100) | 1 | 0
  Titration Period: > 3 RBC Units (n = 89, 100) | 0 | 0
  Evaluation Period: 1 RBC Unit (n = 89, 100) | 1 | 3
  Evaluation Period: 2 RBC Units (n = 89, 100) | 3 | 4
  Evaluation Period: 3 RBC Units (n = 89, 100) | 1 | 2
  Evaluation Period: > 3 RBC Units (n = 89, 100) | 0 | 1
  Safety Follow-up Period: 1 RBC Unit (n = 83, 90) | 0 | 0
  Safety Follow-up Period: 2 RBC Units (n = 83, 90) | 1 | 1
  Safety Follow-up Period: 3 RBC Units (n = 83, 90) | 0 | 0
  Safety Follow-up Period: >3 RBC Units (n = 83, 90) | 0 | 0

ADVERSE EVENTS:
Time Frame: 41 Weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Epoetin Alfa Alternative Titration | Epoetin Alfa USPI Titration
Serious Adverse Events (participants affected / at risk) | 37/104 | 39/107
Other Adverse Events (participants affected / at risk) | 19/104 | 26/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa Alternative Titration (N=104) | Epoetin Alfa USPI Titration (N=107)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 2
Cardiac valve disease (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis escherichia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 6
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 3 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 4
Encephalopathy (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
End stage renal disease (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Steal syndrome (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa Alternative Titration (N=104) | Epoetin Alfa USPI Titration (N=107)
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 8
Haemoglobin increased (Investigations) | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Hypertension (Vascular disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.